CLINICAL TRIAL: NCT03578250
Title: Upper Extremity Training by Error Augmentation in Post-stroke Individuals
Brief Title: Error Augmentation Training Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHaifa062018
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Stroke
Keywords: Stroke; Error augmentation; Rehabilitation; Cerebellum; Motor learning; Adaptation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Training of the upper extremity on a robotic device. Participants will carry out hand reaching movement for multiple directions in 3 dimensions, while grasping the robotic handle according to assignments given by the robotic device.
  During training the robotic device will apply error augmentation force-field to perturbate the arm of the participant away from the straight trajectory line.
  Interventions: Other: Robotic Training
- Control group (Experimental): Training of the upper extremity on a robotic device. Participants will carry out hand reaching movement for multiple directions in 3 dimensions, while grasping the robotic handle according to assignments given by the robotic device.
  During training the robotic device will not apply any perturbations on the participant's arm.
  Interventions: Other: Robotic Training

INTERVENTIONS:
Other: Robotic Training — Upper extremity training on a robotic device with or without error augmentation force field.

SUMMARY:
Post-stroke individuals continue to suffer from significant motor impairments years after the stroke. Motor recovery is usually limited to the first 6 month after the stroke, in which the majority of improvements occur at the first three months. Error augmentation (EA) training using a robotic apparatus was suggested to enhance motor recovery by exploiting the adaptation mechanisms within the intact cerebellum in individuals who sustained cortical stroke.

The aim of this study is to investigate whether error augmentation training for the upper extremity may enhance motor recovery in individuals that sustained cortical stroke.

Fifty post-stroke individuals will be randomaly assigned into either EA training (study group- SG) or robotic training in null field environment (control group- CG). Both groups will carry out the same treatment protocol on the robotic device in addition to the standard rehabilitation protocol of the rehabilitation center. Treatment protocol will be consisted of about six training sessions on the robotic device, taken twice or three times a week for two to three weeks. Each training session will be composed of 20-30 minutes upper extremity training with or without EA force field.

Motor performance will be evaluated before and after the treatment protocol by the Fugl-Meyer Assessment scale.

DETAILED DESCRIPTION:
Post-stroke individuals continue to suffer from significant motor impairments years after the stroke. Motor recovery is usually limited to the first 6 month after the stroke, in which the majority of improvements occur at the first three months. Error augmentation (EA) training using a robotic apparatus was suggested to enhance motor recovery by exploiting the adaptation mechanisms within the intact cerebellum in individuals who sustained cortical stroke.

The aim of this study is to investigate whether error augmentation training for the upper extremity may enhance motor recovery in individuals that sustained cortical stroke.

Fifty post-stroke individuals will be randomaly assigned into either EA training (study group- SG) or robotic training in null field environment (control group- CG). Both groups will carry out the same treatment protocol on the robotic device in addition to the standard rehabilitation protocol of the rehabilitation center. Treatment protocol will be consisted of about six training sessions on the robotic device, taken twice or three times a week for two to three weeks. Each training session will be composed of 20-30 minutes upper extremity training with or without EA force field.

Motor performance will be evaluated before and after the treatment protocol by the Fugl-Meyer Assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Cortical stroke, unilateral hemiparesis

Exclusion Criteria:

* other neurological disorders (Alzheimer's disease, PD), complete plegia,unilateral neglect,sensory aphasia, Mini Mental State Examination<20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Scale | Baseline
  Clinical test for the assessment of motor impairments of the upper extremity

CONTACTS AND LOCATIONS:
Overall Officials: Eli Carmeli, PhD, Study Director — Professor
Locations (1):
- Bait Balev, Nesher, Israel